CLINICAL TRIAL: NCT00138853
Title: A Roentgen Stereophotogrammetric Analysis on Migration of Knee Prostheses. A Randomised Prospective Study of Tantalum Versus Titanium Implants.
Brief Title: A Roentgen Stereophotogrammetric Analysis on Migration of Knee Prostheses.
Acronym: Ti-Tan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20030119
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
Keywords: RSA; Genoarthrosis; Knee arthroplasty; Micromotion of polyethylene liner
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tantalum knee (Active Comparator): Tantalum Tibial component, uncemented
  Interventions: Device: Tibial component
- Titanium Knee (Active Comparator): Titanium Tibial Component, screw fixed
  Interventions: Device: Tibial component

INTERVENTIONS:
Device: Tibial component — Tibial component inserted at the time of surgery
  Other Names: NexGen Tantalum Tibial Plate; NexGen Titanium Tibial Plate, screw fixed

SUMMARY:
The purpose of this study is to compare the early migration of two uncemented total knee arthroplasties with different metal coating. Only the tibial prosthesis plateau varies. One is made out of tantalum and has two short pegs for fixation into the tibia while the other is covered by titanium fiber-mesh on the bone-near site and has 4 short pegs for screw fixation into the tibia.

DETAILED DESCRIPTION:
Around 4% of total knee arthroplasties (TKA) are revised 15 years after the primary operation, most due to loosening of the implant. The use of uncemented prostheses are expected to extend the fixation time and thereby the years of TKA survival. When a cementless implant is inserted, direct bone ingrowth to the implant depends on a complete primary stabilisation. Movement between the bone and implant will cause a fibrous membrane leading to micromotions. Micromotions can be evaluated by radiophotogrammetric analysis (RSA) in early follow-up and they have been shown to be a prognostic marker for painful loosening of the implant.

Tantalum is a fairly new biomaterial designed with a high and bone-binding porosity. Tantalum has already proven to be a good prosthesis material facilitating fast bone-ingrowth and supplying mechanical qualities in the bone-prosthesis interface that surpasses the qualities of regular prosthesis materials by uncemented method. Titanium on the other hand has been used as a prosthesis coating for years and also promote prosthesis fixation by osteointegration.

The purpose of this study is to compare the early migration of two uncemented total knee implants with different metal coating and fixation method. Only the tibial prosthesis plateau varies in design. One plateau is a 2 pegged tantalum monobloc and the other plateau is a modular titanium fiber-mesh coating with 4 short pegs for screw fixation into the tibia.

Furthermore the extend of the expected micromovements between the polyethylene liner and the metal backing of the titanium plateau will be compared to the stable tantalum monobloc.

Theoretically tantalum should allow a more optimal coating for bone ingrowth, but as primary stability is also important for longterm prostheses survival the method of primary fixation could alså play a role.

To evaluate both the plateau-bone micromotions and the polyethylene-prosthesis micromovements metal markers have been placed on the prosthesis pre-operatively and furthermore into the tibial bone and into the tibial polyethylene during surgery allowing us to evaluate stereo x-rays by a photogrammetric analyses called RSA at the Orthopaedic Center, Aarhus University Hospital. Follow-up stereo x-rays will be scheduled for 1 week, 3 months, 6 month, 1 years, 2 years and 5 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one- or double-sided primary knee arthrosis.
2. Patients with a sufficient bone quality for implantation of an uncemented prosthesis.
3. Informed and written patient consent.

Exclusion Criteria:

1. Patients with neuromuscular or vascular diseases in the affected leg.
2. Patients who peroperatively are estimated unsuitable for an uncemented knee arthroplasty e.g. due to bone cysts or dilution of the bone mass.
3. Patients who use non-steroid anti-inflammatory drugs (NSAID) and cannot refrain from taking them postoperatively (this includes COX-2-inhibitors).
4. Patients with osteoporosis estimated from the preoperative x-ray or former diagnosis of osteoporosis.
5. Patients with fracture sequelae.
6. Women, who are pregnant or are at risk of getting pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Polyethylene wear (mm) of the medial and lateral knee prosthesis compartments at 5 years followup measured with model-based radiostereometry | Up to 5 years

SECONDARY OUTCOMES:
Difference in MPTM (mm) tibial component migration from 2-5 years (stabilization 3) measured with model-based radiostereometry | up to 5 years
Number of implants migrating above 0.2mm MTPM from 1-2 years (stabilization 2) and 2-5 years (stabilization 3) measured with model-based radiostereometry | Up to 5 years
Osteolysis (radiolucent lines >1 mm) in the tibial periprosthetic region measured on radiographs | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD, Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Palle Juul-Jensens Boulevard 165, 8200 Aarhus N, Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital., Aarhus, Denmark